CLINICAL TRIAL: NCT04940715
Title: Efficacy of Passive Joint Mobilization vs Mobilization With Movement on Pain Processing in Patients With Chronic Low Back Pain: a Double-blinded, Randomized Clinical Trial.
Brief Title: Efficacy of Passive Joint Mobilization vs Mobilization With Movement on Pain Processing in Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1003202108421
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic low back pain; Pain processing; Manual Therapy
MeSH Terms: interventions — Movement

STUDY DESIGN:
Intervention Model Description: Parallel assignment. Randomized, longitudinal, experimental, prospective, parallel and double-blind study with chronic low back pain adults.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Passive joint mobilization (Experimental): Patients lay down on a prone position, with their hands around the body and neck placed comfortable. The therapist performed a postero-anterior joint mobilization using Maitland's technique, applying pressure to spinous process of targeted vertebra (the one who reproduces patient's symptoms).
  Interventions: Other: Passive joint mobilization
- Mobilization with movement (Experimental): Patients perform their painful movement (flexion, extension…). If pain wasn't reproduced, a combination of movements will be performed (flexion + rotation…). The most painful vertebral level was assessed too with passive accessory vertebral movements. Afterwards, with the patient on a seated position on a stretcher with feet supported and a belt around the waist, the therapist performed a sustained glide on the targeted vertebra (spinous process) with the force and direction that relieved pain to the lowest level.
  Interventions: Other: Mobilization with movement
- Control group (No Intervention): Patients were measured at baseline and then were placed on "wait list" until the end of the study. At this time, they were measured again.

INTERVENTIONS:
Other: Passive joint mobilization — Dosage: 5 sets of 2 minutes with 30 seconds of rest were applied, with a strong force (>50% of maximum therapist strength), according to patient's irritability and severity.
  Arms: Passive joint mobilization
Other: Mobilization with movement — Dosage: 3 sets of 10 repetitions were performed, with 1-2 minutes of rest between sets.
  Arms: Mobilization with movement

SUMMARY:
Patients with chronic low back pain may have altered pain processing, making them vulnerable to pain or disability. It can be measured with test like pressure pain threshold, temporal summation or conditioned pain modulation. Manual therapy has shown improve this pain processing variables in other conditions (like knee osteoarthritis or lateral elbow pain), although the quality of the evidence is low in terms of temporal summation and controversial in terms of conditioned pain modulation. There are not studies that had investigated the impact of manual therapy techniques on pain processing in patients with chronic low back pain.

DETAILED DESCRIPTION:
Study Aims:

Aim #1: The main objective of this study is to determine the efficacy of two manual therapy approaches (passive joint mobilization and mobilization with movement) on pain (measured with Visual Analogue Scale) and pain processing (measured with pressure pain threshold, temporal summation and conditioned pain modulation) in patients with chronic low back pain and see its results on short, medium and long term.

Aim #2: The secondary objective is to compare the effect of both manual therapy techniques with an inactive control group in terms of pain and pain processing.

Aim #3: Determine the efficacy of manual therapy on intervention groups on psychological outcomes as catastrophizing (Pain Catastrophizing Scale), kinesiophobia (Tampa Scale of Kinesiophobia) and depression (Beck Depressive Inventory) and compare them with control group.

Methodology Research Design: Randomized, longitudinal, experimental, prospective, parallel and double-blind study with patients with chronic low back pain.

Participants: Adults between 18-65 years old residing Comunidad de Madrid, all of whom were recruited personally for the study. All patients will read the information sheet explaining what the study will consist, as well as the informed consent form, which they will sign voluntarily beforehand.

Sample Size: The sample size will be calculated by means of the "Gpower 3.0.18" computer program.

Randomization: Randomization will be done through the GraphPad software (GraphPad Software, Inc CA 92037 USA). Patients who meet the inclusion criteria and have none of the exclusion criteria will be entered into the study and the sample will be randomized to obtain three groups in opaque and sealed envelopes: A (passive joint mobilization), B (mobilization with movement) and C (control group).

Masking: The double-blind criteria are met, in which the subjects participating in the study will not know the group to which they were assigned, as well as the physiotherapist in charge of collecting the outcomes data.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific chronic low back pain patients, without lower limb pain
* Pain lasting 6 months or more
* Pain measure of 2 or more on a 0 to 10 scale
* Age between 18-65 years old
* Haven't received physical therapy during last month

Exclusion Criteria:

* Radiculopathy
* Neurological signs, symptoms or deficit
* Rheumatic/autoimmune/systemic disease
* History of fracture, trauma or previous spinal surgery
* Pregnancy
* Disc herniation
* Neuropathic pain
* Active cancer
* Spondylolysis/Spondylolisthesis
* Cognitive impairment
* Long-term opioid intake

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Pain | Change from baseline, after the first intervention, after the last intervention and at both follow-up (1 month and 3 months) periods.
  Visual Analogue Scale (VAS) was used to measure pain. It consists of a 100mm length line and has written "no pain" and "worst pain imaginable" on its ends and measures pain intensity. The confidence and reliability of this scale has been approved and validated in different studies.
Pressure pain threshold | Time Frame: Change from baseline, after the first intervention, after the last intervention and at both follow-up (1 month and 3 months) periods.
  A digital algometer was used to measure mechanical hyperalgesia. The model was de X® brand, consisting of a 1cm2 cylindrical rubber attached to a pressure gauge, calibrated in kilograms (kg). The scale expressed in kg/cm2 was used. Before the measurement, patients were trained in forearm muscles through a trial session. They were instructed to say STOP when the pressure sensation was painful. For the measurement, patients lay down on prone position on the stretcher and the algometer was placed perpendicular to skin on the measured points, who were marked prior to measurement (2cm lateral to L5 spinous process, C2 spinous process, ipsilateral anterior tibialis and contralateral epicondyle). A rest period of 30 seconds was established between the measurements. For each point, three measurements were done and their mean was calculated and recorded for analysis. The minimum detectable change (CMD) for considering the results as clinically relevant was established at 15% minimum.
Temporal summation | Change from baseline, after the first intervention, after the last intervention and at both follow-up (1 month and 3 months) periods.
  Temporal summation was measured with Von Frey monofilaments. Patients lay down on prone position and measurements were taken 1cm lateral to spinous process of L4. First, a single stimulus was applied and the patient assessed the pain intensity on a 0-10 numeric rating scale. After that, 10 rhythmic stimuli were applied on the same spot (1 stimuli per second) and the patient assessed again the pain intensity. The temporal summation effect was calculated as the difference between the mean rating of the three repetitions of one stimulus and the mean rating of the three repetitions of 10 stimulus.
Conditioned pain modulation | Change from baseline, after the first intervention, after the last intervention and at both follow-up (1 month and 3 months) periods.
  Conditioned pain modulation was measured with tourniquet test. A sphygmomanometer was used to induce ischemic muscle pain as conditioning stimulus (model X®). It was applied around the contralateral upper arm, 3cm proximal to cubital fossa. Now, pressure pain threshold 2cm lateral to L5 spinous process was measured. Afterwards, the cuff was inflated to 260mmHg and maintained until the patient perceived a pain intensity of 6 on a 0-10 numeric rating pain scale. Then, the pressure pain threshold was measured again at the same spot during the conditioning stimulus and then the cuff pressure was released. The conditioned pain modulation value is the result of the subtraction of the value of the PPT during the conditioning stimulus minus the PPT without it.

SECONDARY OUTCOMES:
Pain Catastrophizing | Changes from baseline, after the last intervention and at both follow-up periods (1 month and 3 months).
  Catastrophism was measured with Spanish version of Pain Catastrophizing Scale. It's a 13-item self-report measure of catastrophizing and it's constructs as rumination, magnification and helplessness. It must be answered by numeric values between 0 (not at all) and 4 (all the time), with a maximum score of 52 points. The minimal detectable change was identified at 9.1 points.
Kinesiophobia | Changes from baseline, after the last intervention and at both follow-up periods (1 month and 3 months).
  Fear of movement was measured with Spanish version of Tampa Scale of Kinesiophobia. It's an 11-item self-report questionnaire to assess fear of movement-related pain. It's divided on two subscales, one related to Fear of Activity and the other related to Fear of Harm. The score ranges between 11-44 points, with higher scores associated with greater kinesiophobia. The minimal detectable change score was 5.6.
Depression | Changes from baseline, after the last intervention and at both follow-up periods (1 month and 3 months).
  Depressive symptoms were measured with Spanish version of Beck Depressive Inventory. It's a 21-item self-report questionnaire to identify symptoms associated with depression. Each question has a value between 0-3 points, in terms of intensity. The questionnaire assesses cognitive, affective and neurovegetative depressive symptoms, with total score range from 0 to 63.
Central sensitization | Changes from baseline, after the last intervention and at both follow-up periods (1 month and 3 months).
  Central sensitization was measured with Spanish version of Central Sensitization Inventory. This inventory tries to identify the presence of central sensitization. Part A of the questionnaire assess 25 health-related symptoms that are common to central sensitization, with total score ranging from 0 to 100. Part B (not scored) asks about specific disorders or pathologies associated with central sensitization.
Disability | Changes from baseline, after the last intervention and at both follow-up periods (1 month and 3 months).
  Disability was measured with Spanish version of Oswestry Disability Index. This tool assess pain-related disability in people with low back pain. This index assess 1 item on pain and 9 items on activities of daily living (personal care, lifting, walking…). Scores ranges from 0 (no disability) to 100 (maximum disability).

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Martínez Pozas, PhD candidate, Principal Investigator — Universidad Rey Juan Carlos (Madrid); Eleuterio A. Sánchez Romero, PhD, Study Director — Universidad Europea de Madrid (Madrid); Josué Fernández Carnero, PhD, Study Director — Universidad Rey Juan Carlos (Madrid); Héctor Beltrán Alacreu, PhD, Study Director — Universidad de Castilla La-Mancha (Toledo)
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] den Bandt HL, Paulis WD, Beckwee D, Ickmans K, Nijs J, Voogt L. Pain Mechanisms in Low Back Pain: A Systematic Review With Meta-analysis of Mechanical Quantitative Sensory Testing Outcomes in People With Nonspecific Low Back Pain. J Orthop Sports Phys Ther. 2019 Oct;49(10):698-715. doi: 10.2519/jospt.2019.8876. Epub 2019 Aug 23. PMID 31443625
- [Background] Neelapala YVR, Bhagat M, Frey-Law L. Conditioned Pain Modulation in Chronic Low Back Pain: A Systematic Review of Literature. Clin J Pain. 2020 Feb;36(2):135-141. doi: 10.1097/AJP.0000000000000778. PMID 31764164
- [Background] McPhee ME, Vaegter HB, Graven-Nielsen T. Alterations in pronociceptive and antinociceptive mechanisms in patients with low back pain: a systematic review with meta-analysis. Pain. 2020 Mar;161(3):464-475. doi: 10.1097/j.pain.0000000000001737. PMID 32049888
- [Background] Alkhawajah HA, Alshami AM. The effect of mobilization with movement on pain and function in patients with knee osteoarthritis: a randomized double-blind controlled trial. BMC Musculoskelet Disord. 2019 Oct 18;20(1):452. doi: 10.1186/s12891-019-2841-4. PMID 31627723
- [Background] Lascurain-Aguirrebena I, Newham D, Critchley DJ. Mechanism of Action of Spinal Mobilizations: A Systematic Review. Spine (Phila Pa 1976). 2016 Jan;41(2):159-72. doi: 10.1097/BRS.0000000000001151. PMID 26751060
- [Background] Aspinall SL, Jacques A, Leboeuf-Yde C, Etherington SJ, Walker BF. No difference in pressure pain threshold and temporal summation after lumbar spinal manipulation compared to sham: A randomised controlled trial in adults with low back pain. Musculoskelet Sci Pract. 2019 Oct;43:18-25. doi: 10.1016/j.msksp.2019.05.011. Epub 2019 May 31. PMID 31176287
- [Background] Arribas-Romano A, Fernandez-Carnero J, Molina-Rueda F, Angulo-Diaz-Parreno S, Navarro-Santana MJ. Efficacy of Physical Therapy on Nociceptive Pain Processing Alterations in Patients with Chronic Musculoskeletal Pain: A Systematic Review and Meta-analysis. Pain Med. 2020 Oct 1;21(10):2502-2517. doi: 10.1093/pm/pnz366. PMID 32100027